CLINICAL TRIAL: NCT04933656
Title: Use of Stable Carbon And Nitrogen Isotopes to Improve Dietary Assessment for Cardiovascular Disease
Acronym: I-CAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not renewed.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cheryl A. Anderson, MPH, PhD, Professor, Interim Chair, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16IRG27770080
Record Dates: First submitted 2020-02-21; First posted 2021-06-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adults
Keywords: Isotopes; Sugar; Diet; Health
MeSH Terms: interventions — Floors and Floorcoverings

STUDY DESIGN:
Intervention Model Description: Dietary intervention consisting of four 24-hour feeding periods (1 feeding period per week for 4 weeks).
Who Masked: Participant, Care Provider
Masking Description: Double blinding: Participant and person collecting data measurement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 50g added sugar (Experimental): Crossover design and each participant receives all 4 experimental arms/doses in random order
  Interventions: Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level
- 90g added sugar (Experimental): Crossover design and each participant receives all 4 experimental arms/doses in random order
  Interventions: Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + one serving sugar sweetened beverage
- 130g added sugar (Experimental): Crossover design and each participant receives all 4 experimental arms/doses in random order
  Interventions: Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + two servings sugar sweetened beverage
- 170g added sugar (Experimental): Crossover design and each participant receives all 4 experimental arms/doses in random order
  Interventions: Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + three serving sugar sweetened beverage

INTERVENTIONS:
Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level — 50g added sugar
  Arms: 50g added sugar
Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + one serving sugar sweetened beverage — 90 grams added sugar
  Arms: 90g added sugar
Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + two servings sugar sweetened beverage — 130 grams added sugar
  Arms: 130g added sugar
Dietary Supplement: one 24 hr cycle of meals at a 2000 kcal level + three serving sugar sweetened beverage — 170 grams added sugar
  Arms: 170g added sugar

SUMMARY:
In this research study, the investigators will use a novel approach to measure what people eat. The goal is to find out whether stable isotopes that can be measured in blood, hair, and fingernails are better at measuring what people eat than the surveys that are currently used. To meet the goal, the investigators will do three things. First, the investigators will feed study participants known amounts of foods and nutrients. Second, after study participants have eaten the food, the investigators will measure stable isotopes in samples of study participants' blood, hair, and fingernails. Third, the investigators will determine how well these samples reflect what was eaten. The investigators will also give surveys to study participants to determine how well the surveys reflect what was eaten. This will allow the investigators to do a relative comparison of the measurements from isotopes and surveys.

DETAILED DESCRIPTION:
This is a controlled feeding study in which the relative validity of stable carbon and nitrogen isotope ratio analysis as a biomarker of dietary intake is compared to controlled feedings and multiple 24-hour recalls. Participants will be randomly assigned to a sequence of diets to be fed on four occasions. Participants will undergo 24 hours of controlled feeding on four non-consecutive days over a month-long period. On the day after feeding, participants will complete 24-hour dietary recalls, and provide blood, hair, and fingernail samples for isotope ratio analyses. The investigators will use a crossover design and the diets will be either high or low in C4 plants (i.e., corn and cane products). A 24-hour urine collection will be done at home during each 24-hour feeding period. Participants will have height and weight measured at the screening visit. Weight will also be measured at each study visit. Additionally, data will be collected via questionnaires administered at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* men and women;
* aged 21 and 74 years;
* no history of chronic disease and in general good health;
* able to provide primary study outcome; and
* willing to tolerate study diets designed for controlled feeding.

Exclusion Criteria:

* recent dietary changes, restrictions, allergies or preferences;
* health conditions that require management beyond the scope of the study (e.g. heart failure, kidney disease, liver disease, gastrointestinal disorder);
* history of drug or alcohol abuse;
* plans to leave the San Diego area before study completion; and
* lack of suitability per investigators' discretion.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Carbon isotope values from blood | 30 days
  The ratio of carbon 13 to carbon 12 in human blood will be determined.

SECONDARY OUTCOMES:
Carbon isotope values from hair | 30 days
  The ratio of carbon 13 to carbon 12 in human hair samples will be determined.
Carbon isotope values from fingernails | 30 days
  The ratio of carbon 13 to carbon 12 in human fingernail samples will be determined.
Nitrogen isotope values from blood | 30 days
  The ratio of nitrogen-15 to nitrogen 14 in human blood will be determined.
Nitrogen isotope values from hair | 30 days
  The ratio of nitrogen-15 to nitrogen 14 in human hair will be determined.
Nitrogen isotope values from fingernails | 30 days
  The ratio of nitrogen-15 to nitrogen 14 in human fingernails will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A. Anderson, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States